CLINICAL TRIAL: NCT04088994
Title: Rehabilitation of Hemiplegic Cerebral Palsy Children: Role of Motor Activity and Action Observation Therapy in the Recovery of the Affected Upper Limb
Brief Title: Action Observation Based Rehabilitation of Children With Unilateral Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEREBRALPALSYc1
Record Dates: First submitted 2019-06-13; First posted 2019-09-13 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2021-09

CONDITIONS: Hemiplegic Cerebral Palsy; Motor Activity
Keywords: Hemiplegic Cerebral Palsy; Mirror neuron System; Action Observation; Rehabilitation; fMRI
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental study, with 1:1 allocation ratio and two-armed blind assessment. Randomization will be stratified by age and level of HFC system to obtain two groups balanced with respect to the level of functional impairment of the upper limbs to be subjected to treatment in the two groups. Clinical evaluations will be performed before treatment (T0), at the end of treatment (T1), from 8 to 12 weeks after the end of treatment (T2) and finally, from 24 to 28 weeks after the end of treatment (T3).
  Evaluation by fMRI will be performed at T0 and T1.
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pathological model (Experimental): The children assigned to the experimental group will participate in a rehabilitative protocol based on the AOT observing unimanual and bimanual actions performed by a model with a similar manipulation strategy but improved with respect to the child's current abilities.
  Interventions: Other: AOT Pathological Model Experimental Group
- Healthy model (Active Comparator): The children assigned to the control group will participate in a rehabilitative protocol based on the AOT observing unimanual and bimanual actions performed by a healthy model
  Interventions: Other: AOT Healthy Model Control Group

INTERVENTIONS:
Other: AOT Pathological Model Experimental Group — The children will participate in a rehabilitation intervention based on the observation of unimanual and bimanual actions performed by a model with the same degree of motor impairment, but an improvement on the participant's current abilities.
  Other Names: Pathological Model
  Arms: pathological model
Other: AOT Healthy Model Control Group — The children assigned to the healthy group will participate in a rehabilitative protocol based on the AOT observing unimanual and bimanual actions performed by a healthy model
  Other Names: Healthy Model
  Arms: Healthy model

SUMMARY:
Recent evidence suggested that Action Observation Therapy (AOT), based on observation of actions followed by immediate reproduction, could be a useful rehabilitative strategy for promoting functional recovery of children affected by Unilateral Cerebral Palsy (UCP).

The AOT is based on the discovery of mirror neurons, a class of visuomotor neurons that are activated when the individual performs a targeted action, both when observing the same action performed by another individual.

An important assumption of AOT is that the mirror system, thanks to its visuomotor properties, is able to coordinate visual information with the observer's motor experience. Indeed, the actions outside the individual's behavioral repertoire are elaborated and categorized only on the basis of visual characteristics, without inducing any phenomenon of motor resonance in the observer's brain.

Therefore, given the deficiency of their motor repertoire, children affected by UCP could have a reduced activation of the mirror system during the observation of actions performed by healthy subjects. Nevertheless, this activation could increase during the observation of the same actions performed by a subject with similar motor strategies, due to a similar form of hemiplegia.

The present project is a randomized controlled clinical trial to verify the influence of the observed model on the effectiveness of AOT in the rehabilitation of the affected upper limb in children with UCP. In particular, the study will verify whether the rehabilitation through AOT based on a pathological model (improving the patient's current abilities) gives more results than AOT based on a typical (healthy) development model, as reported by all the documented researches in literature.

Furthermore, to investigate the functional reorganization of the sensorimotor system after rehabilitative treatment, a subgroup of participants will be subjected to a fMRI session (Functional Magnetic Resonance), to verify functional changes, comparing data before and after AOT.

DETAILED DESCRIPTION:
The study will compare two rehabilitation models through AOT to assess feasibility and effectiveness. In the preliminary phase of the study a single rehabilitation treatment protocol will be planned, based on the observation and execution of unimanual and bimanual actions integrated in activities that are significant for the subject's age group. The recorded actions will be performed by a child with typical development and by two hemiplegic children:

1. upper limb disability with grades between 4-5 according to House Functional Classification (HFC) system (corresponding to synergic hand of Ferrari and Cioni's Kinematic Hand Classification).
2. upper limb disability with grades between 6-7 according to HFC system (corresponding to subfunctional hand of Ferrari and Cioni's Kinematic Hand Classification).

The participants (N. 26) randomly assigned to the experimental group will be subjected to the rehabilitation protocol through AOT based on the observation of the "Pathological Model". The model, while showing a manipulation strategy similar to that of the study participant, will show an improvement with respect to the patient's current abilities. The children randomly assigned to the control group will be subjected to the rehabilitation treatment protocol through AOT based on the "Typical developmental model".

Both experimental and control treatment will consist of a minimum of 10 hours (min. 10, max 15) for a period of 15 consecutive working days (3 weeks). Each video sequence will show a specific action repeated several times for 3 minutes. Subsequently, participants will be asked to perform the action observed with their hemiplegic upper limb or with both upper limbs for a maximum of 3 repetitions.

A subgroup of study participants (N. 8+8) from both groups will undergo two fMRI sessions, before and immediately after the AOT.

The fMRI session consists of two experimental tasks:

1. action observation (functional session 1-2), in which patients will observe short videos in which actions are performed with the right hand from a subjective perspective.
2. motor task (session 3), in which actions consist in reaching-grasping an object (a cube, a sphere or a cylinder) and putting it into boxes, placed on the right and on the left of the object.

The study consists of two experimental conditions:

1. Observation of the paretic hand, in which the actions will be performed by another patient with UCP.
2. Observation of the healthy hand, in which the action will be reproduced by a healthy model.

The aim of the study is to investigate the functional reorganization of sensorimotor system comparing functional activation before and after rehabilitation with AOT.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of UCP according to definition (MRI and clinical history)
* age 6-16 years at the time of recruitment;
* mild or moderate disability of the upper limb: score between 4 and 7 according to the House Functional Classification (HFC) system;
* sufficient cooperation and understanding to participate in the activities, according to the doctor/physiotherapist who is treating the child and to the neuropsychological evaluation.

Exclusion Criteria:

* cognitive, visual or auditory impairments;
* history of seizures or seizures not well controlled by therapy;
* upper limb surgery within 8 months prior to enrollment;
* upper limb botulinum toxin injection (BoNT-A) within 6 months prior to enrollment.

Additional exclusion criteria for participants in fMRI sessions:

* insufficient cooperation to participation in neuroimaging studies lasting about 30 minutes;
* presence of contraindications to instrumental investigations using 3 Tesla Magnetic Resonance system (implants, metal prostheses, shunts etc.). The presence of these contraindications will be verified by the use of a preliminary questionnaire administered to the parents.
* < 9 years at the time of recruitment.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Change in Assisting Hand Assessment (AHA) | Change from baseline (T0) AHA score to the end of the 3 weeks of treatment (T1), at 8 to 12 weeks (T2) and at 24 to 28 weeks (T3) follow up.
  The AHA measures the effectiveness with which a child with unilateral upper limb disabilities use their affected hand in the bimanual activity with a total raw score range between 22-88 points (the rating scale categories is: 4=effective, 3=somewhat effective, 2=ineffective, and 1=does not do). The higher score indicating higher ability.

SECONDARY OUTCOMES:
Change in Melbourne Assessment of Unilateral Upper Limb Function (MUUL) | Change from baseline (T0) MUUL score to the end of the 3 weeks of treatment (T1), at 8 to 12 weeks (T2) and at 24 to 28 weeks (T3) follow up.
  MUUL is a measure of the unilateral upper limb function. It consists of 16 items that include: reaching, grasping, releasing, manipulating, which estimates 4 domains of movement quality (range, accuracy, fluidity, dexterity). A score from 0 to 3 or 4 is assigned for each domain. Higher scores are associated with better performances.
Change in Ability Hand Kids questionnaire (ABILHAND-Kids) | Change from baseline (T0) ABILHAND-Kids score to the end of the 3 weeks of treatment (T1), at 8 to 12 weeks (T2) and at 24 to 28 weeks (T3) follow up.
  The ABILHAND-Kids is a measure of bimanual performance in activities of daily living.The scale measures a person's ability to manage daily activities that require the use of the upper limbs.The total score based on 21 activities. The parent is asked to rate his/her perception on the response scale as "Impossible", "Difficult" or "Easy" (0 = "Impossible", 1 = "Difficult" or 2 = "Easy").The total score based on 21 activities is then converted into a linear measure of manual ability (logits).
Change in Activities Scale for Kids-Performance Version (ASKp) | Change from baseline (T0) ASKp score to the end of the 3 weeks of treatment (T1), at 8 to 12 weeks (T2) and at 24 to 28 weeks (T3) follow up.
  The ASKp measure physical function and disability in children with musculoskeletal disorders based on their perspective of what they have been doing at home, at school, and on the playground. ASKp is a child self-report questionnaire, which can be parent-reported if necessary. Scale ranges from 0 to 100 with higher scores representing more physical activity.
Change from baseline of functional magnetic resonance imaging (fMRI) analysis | Baseline (T0), T1 (at the end of the 3 weeks of treatment)
  fMRI action observation task

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Fogassi, PhD, Principal Investigator — University of Parma
Locations (1):
- IRCCS S. Maria Nuova Hospital - Rehabilitation unit for severe disabilities in the developmental age, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No
Derived data supporting the findings of this study will be available from the corresponding author upon reasonable request.

REFERENCES:
- [Result] Errante A, Di Cesare G, Pinardi C, Fasano F, Sghedoni S, Costi S, Ferrari A, Fogassi L. Mirror Neuron System Activation in Children With Unilateral Cerebral Palsy During Observation of Actions Performed by a Pathological Model. Neurorehabil Neural Repair. 2019 Jun;33(6):419-431. doi: 10.1177/1545968319847964. Epub 2019 May 10. PMID 31072215
- [Result] Bressi B. Modulating the motor system by action observation in right hemiplegic cerebral palsy: an fMRI study. Nov. 2016, BSc Thesis in Physical Therapy. University of Modena and Reggio Emilia, Italy.